CLINICAL TRIAL: NCT00001238
Title: Von Hippel-Lindau (VHL): Clinical Manifestations, Diagnosis, Management and Molecular Bases of Inherited Renal and Other Urologic Malignant Disorders
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890086; 89-C-0086; NCT00019617 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Kidney Cancer; Urologic Malignant Disorders; Renal Cell Carcinoma; Familial Renal Cancer (FRC); Clear Cell Renal Cancer
Keywords: Hereditary Papillary Renal Cancer (HPRC); Birt Hogg Dube (BHD); Hereditary Leiomyomatosis and Renal Cell Carcinoma (HLRCC); Pheochromocytoma; Von Hippel-Lindau (VHL)
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Hereditary leiomyomatosis and renal cell cancer; Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Disease Category I: Individuals, biologic family members with a suspected or an established diagnosis of an inherited urologic malignancy in which the disease gene is known, including VHL and HPRC
- Disease Category II: Individuals and biologic family members with a suspected or an established diagnosis of an inherited urologic malignancy in which the disease gene is not yet known
- Disease Category III: Individuals and biologic family members with a urologic malignant disease of suspected, but not proven genetic etiology

SUMMARY:
We will investigate the clinical manifestations and molecular genetic defects of heritable urologic malignant disorders. Families with urologic malignancy with known or suspected genetic basis will be enrolled. Affected individuals or individuals suspected of having a germline urologic malignant disorder will undergo periodic clinical assessment and genetic analyses for the purpose of: 1) definition and characterization of phenotype, 2) determination of the natural history of the disorder, and 3) genotype/phenotype correlation. Genetic linkage studies may be performed in situations in which the genetic basis of the disorder has not been elucidated.

...

DETAILED DESCRIPTION:
Background:

* Disorders under investigation are: Autosomal dominant inherited urologic malignant disorders including: von Hippel-Lindau (VHL), hereditary papillary renal cancer (HPRC), Birt Hogg Dube (BHD) and hereditary leiomyomatosis and renal cell carcinoma (HLRCC) as well as familial renal cancer.
* Studies have led to the identification and characterization of the VHL, HPRC, FLCN and HLRCC genes.
* The genetic etiology of the most common type of inherited kidney cancer, familial renal cancer (FRC), remains to be determined.

Objectives:

* To characterize the natural and clinical histories of inherited urologic malignant disorders.
* To determine the genetic etiology of hereditary urologic malignant disorders in which the gene variation is unknown, by linkage analysis, positional cloning and evaluation of candidate genes.
* To correlate specific mutations and their associated protein domains with disease phenotypic expression based on parameters including presenting age, clinical manifestations, histopathology and rate of recurrence.
* To identify and describe as yet unknown or uncharacterized inherited urologic malignant disorders.

Eligibility:

* Individuals and biologic family members with a suspected or an established diagnosis of an inherited urologic malignancy in which the disease gene is known, including von Hippel-Lindau (VHL) and hereditary papillary renal carcinoma (HPRC).
* Individuals and biologic family members with a suspected or an established diagnosis of an inherited urologic malignancy in which the disease gene is not yet known, specifically hereditary forms of Type II papillary renal cancer, clear cell renal carcinoma, renal oncocytoma, chromophobe renal carcinoma or Birt Hogg Dube.
* Individuals and biologic family members who have urologic malignant diseases of suspected, but not proven genetic etiology, including families with more than one individual affected by the same or related cancers.

Design:

* These rare families will be recruited to genetically confirm diagnosis, determine size and location of renal tumors, size at presentation, growth rate and metastatic potential of renal tumors.
* Genetic testing will be offered to gain appreciation of the effect of mutations on the relative activity of various germline and somatic mutations.
* We will determine if there is a relationship between mutation and disease manifestations and phenotype.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must be greater than or equal to 2 years of age. All participants and guardians (for children younger than 18 years of age) must sign an informed consent document indicating their understanding of the investigational nature and the risks of this study before any protocol related studies are performed.

Criteria for Acceptance into this Study (i.e., Disease Categories):

Disease Category I

Individuals and biologic family members with a suspected or an established diagnosis of an inherited urologic malignancy in which the disease gene is known, including von Hippel-Lindau (VHL) and hereditary papillary renal carcinoma (HPRC).

Disease Category II

Individuals and biologic family members with a suspected or an established diagnosis of an inherited urologic malignancy in which the disease gene is not yet known, specifically hereditary forms of Type II papillary renal cancer, clear cell renal carcinoma, renal oncocytoma, chromophobe renal carcinoma or Birt Hogg Dube.

Disease Category III

Individuals and biologic family members who have urologic malignant diseases of suspected, but not proven genetic etiology, including families with more than one individual affected by the same or related cancers. A total of 5000 individuals will be enrolled during the study (i.e., that includes individuals registered since the beginning of the protocols in 1989 (89C0086) and 1999 (99C0101)).

Enrollment per Subject Category (to include both affected and unaffected biologic relatives)

Subject Category A:

Category A will include individuals, and biologic relatives, who may or may not be affected who will be evaluated in the Warren G. Magnuson Clinical Center. Individuals in this category will be eligible if they or their biologic family members manifest one or more of the following features in a pattern suggestive of a heritable urologic malignant disorder:

* One or more histologically proven or suspected renal carcinomas and/or cysts
* Cerebellar, spinal, medullary or cerebral hemangioblastomas
* Retinal angioma
* Pancreatic neuro-endocrine carcinoma,micro cystadenoma and/or cysts
* Pheochromocytoma
* Papillary cystadenoma of the epididymis or broad ligament
* Endolymphatic sac tumor
* Cutaneous fibrofolliculomas or multiple skin-colored papules
* History of spontaneous pneumothorax
* Lung cysts
* Thyroid carcinoma
* Intestinal polyposis plus/minus colon cancer
* Cutaneous or Uterine leiomyoma or uterine leiomyosarcoma, sarcoma

Subject Category B:

Category B will include individuals and the biologic relatives of patients with inherited urologic malignancies with the above listed clinical findings who live at a distance and who will not be evaluated at the Clinical Center. In some cases, local diagnostic testing may be necessary for these individuals in addition to collection of a blood sample for molecular analysis.

Subject Category C:

Category C will include biologic relatives who enroll in this study primarily for genetic linkage studies. These individuals will contribute a blood sample for DNA analysis only. No imaging diagnostic testing will be performed on individuals from this category.

EXCLUSION CRITERIA:

None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with known or suspected inherited urologic malignant disorders and their biologic family members with inherited urologic malignancies will be recruited primarily from the urology, oncology, and genetics communities worldwide
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1990-12-05 (Actual)

PRIMARY OUTCOMES:
Identify and describe as yet unknown or uncharacterized inherited urologic malignant disorders. | on-going
  Collection of blood, tissue & urine to address further scientific questions related to this protocol.
Determine the genetic etiology of hereditary urologic malignant disorders in which the gene variation is unknown, by linkage analysis, positional cloning and evaluation of candidate genes. | on-going
  Collection of blood, tissue & urine to address further scientific questions related to this protocol.
Correlate specific mutations and their associated protein domains with disease phenotypic expression based on parameters including presenting age, clinical manifestations, histopathology and rate of recurrence. | on-going
  Collection of blood, tissue & urine to address further scientific questions related to this protocol.
Characterize the natural and clinical histories of inherited urologic malignant disorders. | on-going
  Collection of blood, tissue & urine to address further scientific questions related to this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: W. Marston Linehan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1989-C-0086.html